CLINICAL TRIAL: NCT05562180
Title: FOOD PRESCRIPTION APP TO EXTEND AND CUSTOMIZE HEALTHY MEALS FOR A BETTER DIET
Brief Title: FOOD PRESCRIPTION APP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Deborah A Cohen, Research Scientist, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3P50MD017344-02S1 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): These participants will use the app to customize their weekly meal plan and grocery delivery
  Interventions: Behavioral: Customized meal plan and grocery delivery
- comparison (No Intervention): These participants will not receive a weekly meal plan and will not get grocery delivery

INTERVENTIONS:
Behavioral: Customized meal plan and grocery delivery — Participants will use an app to customize their meal plans
  Arms: Intervention arm

SUMMARY:
This study will develop and test and app that will create meal plans to improve diet quality and support weight loss. This app will allow participants to customize their meal plans and substitute recipes for nutritionally equivalent options that they find more appealing, thus potentially increasing adherence.

DETAILED DESCRIPTION:
We are specifically planning app to create meal plans that are affordable, meet the recommended dietary allowances (RDAs) and adhere to sustainability guidelines to reduce the food-related carbon footprint. The app will enable participants to customize their weekly meal plans. We hypothesize that having the ability to customize the weekly menus through a FoodRx app will improve outcomes, as the lack of customization appeared to be a barrier for some families to improve their diet quality and achieve weight loss goals. (eg, some families did not like tofu or oatmeal, and would have preferred a substitute). We will be able to test the impact of the Food Rx app by comparing participants who use it to our control group that does not currently have access to the standard menus/grocery delivery or FoodRx app.

ELIGIBILITY:
Inclusion Criteria:

Already enrolled in FoodRx study >18 years BMI>27 and wants to lose weight -

Exclusion Criteria:

Not enrolled in Food Rx

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dietary Quality | 1 month
  HEI (Healthy Eating Index)

SECONDARY OUTCOMES:
weight loss | 1 month
  BMI will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No